CLINICAL TRIAL: NCT00000748
Title: A Randomized, Comparative, Prospective Study of Daily Trimethoprim / Sulfamethoxazole (TMS) and Thrice-Weekly TMS for Prophylaxis Against PCP in HIV-Infected Patients
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Collaborators: Glaxo Wellcome (Industry)
Responsible Party: Sponsor
Model: Parallel | Purpose: Treatment
Other Study IDs: CPCRA 006; 11558 (Registry Identifier: DAIDS ES Registry Number)
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2021-11-04 (Actual); Status verified 2021-10

CONDITIONS: Pneumonia, Pneumocystis Carinii; HIV Infections
Keywords: Trimethoprim-Sulfamethoxazole Combination; Pneumonia, Pneumocystis carinii; Acquired Immunodeficiency Syndrome; AIDS-Related Complex; Sulfamethoxazole-Trimethoprim
MeSH Terms: conditions — Pneumonia, Pneumocystis; HIV Infections; Acquired Immunodeficiency Syndrome; AIDS-Related Complex | interventions — Trimethoprim, Sulfamethoxazole Drug Combination

INTERVENTIONS:
Drug: Sulfamethoxazole-Trimethoprim

SUMMARY:
To compare the safety and efficacy of two dosage regimens (daily and thrice-weekly) of sulfamethoxazole/trimethoprim (SMX/TMP; TMS) in the prevention of Pneumocystis carinii pneumonia (PCP) in high-risk HIV-infected patients.

Previous tests have shown that SMX/TMP given daily is effective in preventing recurrence of PCP and may be effective in preventing PCP in patients who have never developed it. Because SMX/TMP can cause side effects, this study will attempt to determine the safest and most effective dose of this combination.

DETAILED DESCRIPTION:
Previous tests have shown that SMX/TMP given daily is effective in preventing recurrence of PCP and may be effective in preventing PCP in patients who have never developed it. Because SMX/TMP can cause side effects, this study will attempt to determine the safest and most effective dose of this combination.

Patients receive SMX/TMP orally on a daily or thrice-weekly basis. Patients are clinically evaluated every 4 months. Patients on daily SMX/TMP who develop a drug-related toxicity may be switched to thrice-weekly SMX/TMP. Duration of follow-up is 12 months.

ELIGIBILITY:
Inclusion Criteria

Patients must have:

* HIV infection.
* CD4 count <= 200 cells/mm3 OR a history of prior PCP.
* No active pneumocystosis. Patients or their guardians must sign informed consent. Pregnant patients are eligible at the clinician's discretion. Patients who do not meet required laboratory values may be eligible at the discretion of the clinician.

Exclusion Criteria

Co-existing Condition:

Patients with the following symptoms and conditions are excluded:

* Known treatment-limiting reaction to sulfonamides or trimethoprim.

Concurrent Medication:

Excluded:

* Other PCP prophylaxis or medication with anti-PCP activity.

Min Age: 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 2500
Dates: Study Completion 1996-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: W El-Sadr, Study Chair; R Luskin-Hawk, Study Chair
Locations (24):
- United States (24):
  - Community Consortium of San Francisco, San Francisco, California
  - Stanford Univ School of Medicine, Stanford, California
  - Denver CPCRA / Denver Public Hlth, Denver, Colorado
  - Wilmington Hosp / Med Ctr of Delaware, Wilmington, Delaware
  - Veterans Administration Med Ctr / Regional AIDS Program, Washington D.C., District of Columbia
  - AIDS Research Consortium of Atlanta, Atlanta, Georgia
  - AIDS Research Alliance - Chicago, Chicago, Illinois
  - Louisiana Comm AIDS Rsch Prog / Tulane Univ Med, New Orleans, Louisiana
  - Baltimore Trials, Baltimore, Maryland
  - Univ of Maryland at Baltimore, Baltimore, Maryland
  - Comprehensive AIDS Alliance of Detroit, Detroit, Michigan
  - Henry Ford Hosp, Detroit, Michigan
  - Southern New Jersey AIDS Cln Trials / Dept of Med, Camden, New Jersey
  - North Jersey Community Research Initiative, Newark, New Jersey
  - Partners Research, Albuquerque, New Mexico
  - Univ Hosp / HIV - ID Clinic, Albuquerque, New Mexico
  - Addiction Research and Treatment Corp, Brooklyn, New York
  - Clinical Directors Network of Region II, New York, New York
  - Harlem AIDS Treatment Group / Harlem Hosp Ctr, New York, New York
  - Bronx Lebanon Hosp Ctr, The Bronx, New York
  - Portland Veterans Adm Med Ctr / Rsch & Education Grp, Portland, Oregon
  - Philadelphia FIGHT, Philadelphia, Pennsylvania
  - Richmond AIDS Consortium, Richmond, Virginia
  - Univ of Washington / Pacific Med Ctr, Seattle, Washington

REFERENCES:
- [Background] Simon PM, Morse EV, Besch L. Barriers to compliance among women co-enrolled in a PCP prophylaxis and compliance protocol. HIV Infect Women Conf. 1995 Feb 22-24:P109
- [Background] El-Sadr WM, Luskin-Hawk R, Yurik TM, Walker J, Abrams D, John SL, Sherer R, Crane L, Labriola A, Caras S, Pulling C, Hafner R. A randomized trial of daily and thrice-weekly trimethoprim-sulfamethoxazole for the prevention of Pneumocystis carinii pneumonia in human immunodeficiency virus-infected persons. Terry Beirn Community Programs for Clinical Research on AIDS (CPCRA). Clin Infect Dis. 1999 Oct;29(4):775-83. doi: 10.1086/520433. PMID 10589887